CLINICAL TRIAL: NCT04004182
Title: Acute Study of Anthocyanin-rich Bilberry and Polyphenol-rich Apple Extracts on Postprandial Glycaemic Response
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Aberdeen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2019/ROW_Berry/3; The Fruit Bar study (Other: Rowett Institute)
Record Dates: First submitted 2019-06-27; First posted 2019-07-01 (Actual); Last update posted 2022-08-24 (Actual); Status verified 2022-08

CONDITIONS: Glucose Intolerance; Glucose Metabolism Disorders
MeSH Terms: conditions — Glucose Intolerance; Glucose Metabolism Disorders

STUDY DESIGN:
Intervention Model Description: This acute intervention study will have a randomised controlled crossover design where the volunteers will return for 4 stand-alone study sessions
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- OGTT session (Active Comparator): Oral Glucose Tolerance test (OGTT)
  Interventions: Dietary Supplement: Fruit bar with addition of polyphenols
- Fruit bar (Active Comparator): Fruit bar Plus Oral Glucose Tolerance test (OGTT)
  Interventions: Dietary Supplement: Fruit bar with addition of polyphenols
- Fruit bar with bilberry (Experimental): Fruit bar with addition of 600 mg bilberry anthocyanins Plus Oral Glucose Tolerance test (OGTT)
  Interventions: Dietary Supplement: Fruit bar with addition of polyphenols
- Fruit bar with bilberry and apple (Experimental): Fruit bar with addition of 600mg bilberry anthocyanins and 1200mg apple polyphenols Plus Oral Glucose Tolerance test (OGTT)
  Interventions: Dietary Supplement: Fruit bar with addition of polyphenols

INTERVENTIONS:
Dietary Supplement: Fruit bar with addition of polyphenols — Fruit bar with addition of 600mg bilberry anthocyanins and 1200mg apple polyphenols

SUMMARY:
Strategies to control chronic postprandial hyperglycaemia by optimizing the functionality of foods would strengthen efforts to reduce the risk of developing T2D in the general population. Polyphenolic constituents, may help to delay starch and disaccharide digestion and glucose absorption following a carbohydrate-containing meal or beverage. In vitro studies suggest that some berry anthocyanins and apple polyphenols are effective inhibitors of digestive enzymes, α-amylases and α-glucosidases. Furthermore, polyphenols found in berries and apples inhibit the action of intestinal glucose transporters. Human data is limited; however, randomized controlled trials (RCTs) have shown that berries and apple products reduced postprandial glucose concentrations following consumption of either starch, glucose or sucrose loads.

The aim of this study is to test the hypothesis that consumption of a fruit bar containing anthocyanin-rich bilberry and polyphenol-rich apple extracts together with a starch and sucrose meal would reduce the postprandial glycemic response.

This study is a randomized cross over study and will aim to recruit 24 overweight (BMI > 25.0), men or post-menopausal women, aged ≥40 and ≤ 70 years who will attend four study sessions. The first study session will be an oral glucose tolerance test (OGTT) and the remaining three will be identical in all respects except for the composition of the fruit bar. Consecutive blood samples will be collected in all 4 study sessions which will be used to measure glucose, insulin, C-peptide, incretins and lipids.

DETAILED DESCRIPTION:
This acute intervention study will have a randomised controlled crossover design where the volunteers will return for 4 stand-alone study sessions. All study procedures will be carried out at the Human Nutrition Unit (HNU) of the Rowett Institute.

The first study session will be an oral glucose tolerance test (OGTT). The remaining three will be intervention sessions which will be identical in all respects except for the composition of the fruit bar. There will have a minimum of 1 week washout period. Volunteers will be asked to consume a low polyphenol diet three days prior to each intervention. To ensure compliance, participants will be provided with a list of 'allowed' and 'excluded' foods as well as food diaries to complete over the three day period. The Fruit bars will be made in the HNU kitchens by trained staff.

Table 1. Study sessions Intervention/Meal

Oral Glucose Tolerance test (OGTT) Fruit bar Plus OGTT Fruit bar with addition of 600 mg bilberry anthocyanins Plus OGTT Fruit bar with addition of 600mg bilberry anthocyanins and 1200mg apple polyphenols Plus OGTT

The glucose load for the OGTT in all sessions will be given as carbohydrate meal consisting of white bread, spread, low-polyphenol jam. (meal: 75g carbohydrate total)

Screening session Once the volunteer expresses interest in the study, they will be invited to attend a screening visit lasting approximately 1 h. Informed consent will be obtained from all participants, ensuring that they have fully understood all the study procedures before continuing. A full eligibility assessment (for assessing inclusion and exclusion criteria) will be carried out following consenting. This will include the completion of a health screening questionnaire, anthropometric measurements (height, weight, BMI,). HbA1c will be measured using finger prick blood samples. Volunteers fulfilling all the criteria and who wish to continue will be accepted into the study.

OGTT and Intervention sessions (study sessions 1-3)

At each session the volunteers will return for 2 visits.

Visit 1: Pre - Study Session Day This session will last approximately 1 hour. Volunteers will arrive at the HNU on the day preceding the study session day for the insertion of the continuous blood glucose monitoring (CGM) sensor (iPro 2, Medtronic Ltd, UK). Upon arrival, their weight will be measured for calculating BMI. Waist circumference and body fat composition using bio-impedance will be also be measured. The CGM records interstitial glucose levels at five minute intervals and provides a detailed picture of glucose fluxes. The CGM monitors are widely used by diabetics to monitor blood glucose fluxes and are designed for self-insertion. Their accuracy and level of data detail has also made them a powerful and widely used research tool. The sensor will be inserted into the subcutaneous fat layer (just below the skin surface) in the belly area by a trained researcher or HNU staff member. Insertion will be carried out using a tailor-made inserter provided with the CGM which causes minimum discomfort. Following stabilisation of the sensor a data acquisition unit will be attached to it. The sensor will be calibrated using a finger prick blood sample. Volunteers will be shown how to calibrate the CGM at home using a standard blood glucose meter and finger prick samples, and instructed on the times when they would have to do so. Wearing the sensor (which is about the size of a £2 coin) causes minimum discomfort to the wearer and does not hinder daily activities (including sleeping and having baths). The volunteers will be provided with a list of foods to consume that evening before each session day. We will ask the volunteer to consume the same meal before each session day. No restrictions will be made on water.

Visit 2: study session day This session will last approximately 4 h. The volunteers will return to the HNU the following morning in an overnight fasted state of approximately 10 h. A cannula will be inserted into a vein in the antecubital fossa at the front of an elbow of the left or right arm and kept patent with sterile saline (0.9% NaCl). Baseline fasted blood (10 mL) samples will be collected into K-EDTA tubes (6 mL serum). The plasma blood collection tubes will also contain DPP-4 inhibitors to preserve incretin hormone integrity. Following baseline sample collection, volunteers will consume the fruit bar and then the carbohydrate meal within 10 min. Periodic blood samples 10 mL will be collected into K-EDTA tubes at 15min, 30min, 45min, 1h, 1.5h, 2h, 2.5h, and 3h post fruit bar/carbohydrate meal consumption.

At the end of the 3 h, the cannula will be removed; volunteers will consume a standardised lunch the CGM sensor will be removed and volunteers will be free to leave the HNU.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men or post-menopausal women
* Aged ≥40 and ≤ 70 years old.
* BMI > 25.0kg/m2
* HbA1c <6.5%

Exclusion Criteria:

Those with any of the following will be excluded from participation:

* Thromboembolic or coagulation disease
* Unregulated thyroid disease
* Kidney disease
* Hepatic disease
* Severe gastrointestinal disorders
* Pulmonary disease (e.g. chronic bronchitis, COPD, pacemaker implant)
* Nut or date allergy
* Alcohol or any other substance abuse
* Eating disorders
* Women who are lactating or breastfeeding, pregnant
* Allergic/intolerant to foods provided in the study
* Alcohol and/or other substance abuse
* Smoking and the use of e-cigarettes
* Physically active at a competitive level (exercising strenuously on a daily basis for long periods of time)

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2019-06-08 (Actual); Primary Completion 2023-03-01 (Estimated); Study Completion 2023-03-01 (Estimated)

PRIMARY OUTCOMES:
Glucose | Over 3 hours post OGTT
  Changes postprandial blood glucose
Insulin | Over 3 hours post OGTT
  Changes postprandial blood glucose

CONTACTS AND LOCATIONS:
Locations (1):
- University of Aberdeen Rowett Institute of Nutrition and Health, Aberdeen, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Initially via publication in journal and then via this site